CLINICAL TRIAL: NCT03170934
Title: The Effectiveness of Psychotherapy Classes in Reducing Suicidal Ideation
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other); Winnipeg Foundation (Unknown)
Responsible Party: Principal Investigator, Natalie Mota, Assistant Professor/Staff Psychologist, University of Manitoba
Other Study IDs: H2017:068
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychotherapy skills class — Rapid access, large-scale, psychotherapy classes that are open format and delivered in lecture style. One class - Managing Difficult Emotions (MDE) - is an 8-session, DBT-informed program. The other class - Mindfulness-Based Cognitive Behavioral Therapy (CBTm) - is a 4-session program.

SUMMARY:
The proposed study will conduct a preliminary investigation of the effectiveness of two different psychotherapy classes at the Mental Health Crisis Response Centre (CRC) in reducing suicidal ideation. One class - Managing Difficult Emotions (MDE) - is an 8-session, Dialectical Behavioral Therapy-informed program that focuses on skills related to increasing tolerance for distress and emotion regulation such that harmful behaviors are reduced. The other class - Mindfulness-Based Cognitive Behavioral Therapy (CBTm) - is a 4-session program that focuses on challenging and changing maladaptive beliefs and behaviors in order to reduce distress. Both classes are delivered in lecture style, PowerPoint format. The investigators will also examine the effectiveness of participation in psychotherapy classes in reducing symptoms of general psychological distress, depression, anxiety, and emotion dysregulation.

DETAILED DESCRIPTION:
Suicide is the ninth leading cause of death in Canada, and rates are exponentially higher among specific sub-populations of Canadians (Statistics Canada, 2015). Worldwide, approximately 800,000 individuals die by suicide each year (WHO, 2016). A number of interventions, such as psychotherapy, have been shown to effectively reduce suicidal thinking and behaviors; however, several factors often impede or delay access to clinical care. In order to reduce suicide, interventions must not only be evidence-based but also readily accessible and perceived as being helpful by patients (Pagura et al., 2009; Turecki & Brent, 2015). Large, lecture-style, skills-based psychotherapy interventions where patients can join at any session can ensure timely access to services while being relatively unintimidating to patients. However, little research to date has examined the effectiveness of such interventions in reducing suicidality.

There is a dire need to develop evidence-based clinical interventions that can be accessed rapidly by individuals during their time of highest need (Brown & Jager-Hyman, 2014). For example, the first few days and weeks following hospital discharge post-suicide attempt represents the period of highest risk for suicide completion, however, a staggering proportion of individuals do not have an outpatient mental health appointment within this timeframe (Glenn et al., 2015; Olfson et al., 2014). Further, studies have often not evaluated the effectiveness of suicide interventions in "real world" settings and where high-risk subgroups of individuals are included (e.g., substance users) and have not consistently used valid and reliable measures of suicidal ideation (Brown & Jager-Hyman, 2014).

The investigators are unaware of any study to date that has examined the effectiveness of rapid access, large-scale, psychotherapy classes in reducing suicidality in a crisis population.

Primary Aim 1: To examine the effectiveness of rapid access, large volume CBT and DBT-informed psychotherapy classes in reducing suicidal ideation among individuals presenting with a mental health crisis.

Hypothesis: The investigators hypothesize that participation in either class will reduce suicidal thinking, and that decreases in suicidal ideation will be greater among those patients completing the total number of classes.

Secondary Aim 2a: To examine the effectiveness of participation in psychotherapy classes in reducing symptoms of general psychological distress, depression, anxiety, and emotion dysregulation.

Hypothesis 2a: The investigators hypothesize that class participation will result in symptom decreases across all outcomes.

Secondary Aim 2b: To identify the sociodemographic and symptom profile(s) of patients benefiting most from psychotherapy classes as well as the characteristics of patients for whom the classes are not helpful.

Hypothesis 2b: The patient profiles deriving the greatest and least psychological benefit (i.e., changes in suicidality and symptoms) from these classes are more exploratory in nature.

Design and Methods

Participants: Patients accessing care for a mental health crisis at the Crisis Response Centre (CRC) or at hospital emergency departments in the city will be referred to the CRC's Urgent Follow-up Intensive Treatment Team (UFITT). The UFITT program is designed to be as inclusive as possible. Referral criteria include: 1) Being 18 years of age or older, 2) the ability to benefit from and participate in large psychotherapy groups (i.e., absence of active psychotic symptoms, ability to understand and read the class material, etc.), 3) not having mental health needs that would be better served by other community resources (e.g., a severe primary substance use disorder, intimate partner violence, etc.), and 4) not being at immediate risk of harming self or others (i.e., patient is safe to return home and to attend an appointment 1-2 weeks after the walk-in visit). Referrals are reviewed for appropriateness by the UFITT team and patients are subsequently invited to attend an information session in order to learn about the follow-up mental health services available. The majority of patients who attend an information session choose to be enrolled in one of the two available psychotherapy classes at the CRC. It is this subpopulation of patients who will be recruited for the proposed study, and we aim to recruit approximately 250 participants. Each participant will receive a $5 Tim Hortons Gift Card as a token of appreciation for their time.

Consent Procedure: Prior to the start of the UFITT information session, the two study coordinators will describe the study to patients, and will inform them that research assistants will be available after patient appointments to meet with those who are interested in participating. Study procedures will be explained in more detail and written informed consent will be obtained following the information session appointment. Participants will additionally be asked if they would be willing to be contacted in the future. Patients who do not consent to participate in the study will receive usual care and follow-up as per UFITT guidelines.

Study Design and Procedures: The proposed study will collect a prospective cohort of patients participating in the psychotherapy classes and will employ a pre-post design.

UFITT patients currently complete a package of widely used, validated measures at the information session in paper and pencil format that assess symptoms in a number of mental health domains. This package of measures will serve as the baseline assessment in the proposed study. Immediately following the information session, patients meet briefly with a CRC staff member to discuss follow-up services and to receive recommendations related to which UFITT psychotherapy class is most likely to benefit them based on their questionnaire scores. Patients choosing to participate in either of the psychotherapy classes are typically provided with an appointment to a class within one week of their information session date. Patients are encouraged to attend psychotherapy classes weekly and at the completion of their last class, are re-administered a subset of the same outcome measures. In the development of the prospective cohort, the investigators will additionally administer the primary outcome measure, the Beck Scale for Suicidal Ideation (Beck & Steer, 1991), to all consenting study participants, which represents a validated and comprehensive assessment of suicidal thinking. In order to understand changes in suicidal ideation among study participants who both complete and 'drop out' from the classes, research assistants will contact those participants who stop attending classes in order to re-administer the measures by telephone. The data collection period will be approximately ten months.

Intervention: Study participants will take part in one of two psychotherapy classes currently ongoing at the CRC. CBTm is a four session (90 minutes per session) introduction to cognitive behavioral skills for managing symptoms of anxiety and depression. The content includes an introduction to mindfulness, challenging maladaptive thoughts, behavioral activation, exposure, managing anger, problem-solving and goal-setting strategies, sleep hygiene, and healthy living guidelines. Managing Difficult Emotions is based on DBT, an intervention developed by Dr. Marsha Linehan (2014). It is an eight session (90 minutes per session) introduction to selected DBT skills related to mindfulness, emotion regulation, distress tolerance, and interpersonal effectiveness. Although both of these classes have been developed to target transdiagnostic psychological distress, several examples related to suicidal ideation and behavior will be used when teaching the skills. Classes are delivered in PowerPoint format, and class sizes typically range from 10 to 25 patients. Sessions have been developed to stand alone, and patients can join either class at any session. Patient participation is encouraged but not required.

Analytic Plan: Data from the hard copy measures will be entered into an electronic database and statistical analyses will be conducted using SPSS v.22. A comprehensive intention-to-treat analysis will examine change in suicidal ideation - the primary outcome - as assessed by the Beck Scale for Suicidal Ideation. These analyses will include all study participants for whom pre-post scores can be obtained, including non-completers of the classes. Type of class (MDE vs. CBTm) and number of sessions attended will additionally be evaluated as predictors of decreases in suicidal ideation. A parallel analysis will be used to examine the effectiveness of class participation in reducing the secondary outcome measures, namely depression, anxiety, general distress, and emotion dysregulation symptoms from the baseline assessment to the last class completed.

Sociodemographic factors (i.e., sex, age, marital status, employment status, level of education), nature of presenting problem at walk-in (e.g., increase in suicidal ideation/behavior, onset of psychosocial stressors, exacerbated trauma-related symptoms, depression/anxiety), and baseline symptoms of depression, anxiety, distress, and emotion dysregulation will be examined as predictors of suicidal ideation at follow-up using linear regression analysis. This analysis will identify the profile of patients who have benefitted the most and the least from psychotherapy classes, and will include both class completers and non-completers. The type and number of classes attended will also be examined in relation to suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Person has been referred to the UFITT program following a mental health crisis
* 18 years of age or older
* Fluent in English
* Ability to understand and read class material
* Ability to independently complete questionnaires
* Has a contact telephone number

Exclusion Criteria:

* Mental health needs better served by other community resources (e.g., a severe primary substance use disorder, intimate partner violence)
* At immediate risk of harming self or others
* Active psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is patients aged 18 years and older who access care at Manitoba's Crisis Response Centre or at a local emergency department and who have been referred to the CRC's UFITT program. Patients who are deemed by CRC staff as potentially benefitting from UFITT programming are asked to attend an Information Session where they are told about crisis follow-up services and in particular, the two psychotherapy classes available. It is those individuals who choose to be enrolled in one of these classes upon attending an Information Session who will be recruited for the proposed study.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Suicidal ideation | Change from baseline (information class) to class completion or drop-out (either at 4 or 8 weeks, depending on the class being completed)
  Current suicidal thinking, as defined by the Beck Scale for Suicidal Ideation

SECONDARY OUTCOMES:
Anxiety symptoms | Change from baseline (information class) to class completion or drop-out (either at 4 or 8 weeks, depending on the class being completed)
  As defined by the Generalized Anxiety Disorder Scale-7 (GAD-7)
Depression symptoms | Change from baseline (information class) to class completion or drop-out (either at 4 or 8 weeks, depending on the class being completed).
  As defined by the Patient Health Questionnaire-9 (PHQ-9)
Emotion regulation difficulties | Change from baseline (information class) to class completion or drop-out (either at 4 or 8 weeks, depending on the class being completed)
  As defined by the Difficulties with Emotion Regulation Scale
General psychological distress | Change from baseline (information class) to class completion or drop-out (either at 4 or 8 weeks, depending on the class being completed)
  As defined by the DSM-5 Cross-cutting Measure

CONTACTS AND LOCATIONS:
Locations (1):
- Crisis Response Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No